CLINICAL TRIAL: NCT05955781
Title: Effects Of Spinal Mobilization With Leg Movement on Pain And Disability in Patients With Lumbar Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/13
Record Dates: First submitted 2023-07-09; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Prallel Group Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: A Single blinded study will be used in which data analyzer will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Spinal Mobilization with Leg Movement (SMWLM) will be given as intervention to experimental group. Participants will be given Hot pack for 15 minutes, TENS for 10 minutes.
  Interventions: Procedure: Spinal Mobilization With Leg Movement; Procedure: Conventional treatment
- Group B (Active Comparator): The patients will be given Spinal mobilization (transverse glide) on the effected spinous process. The total time duration will be 25-30 minutes. Participants will be given Hot pack for 15 minutes, TENS for 10 minutes.
  Interventions: Procedure: Spinal Mobilization; Procedure: Conventional treatment

INTERVENTIONS:
Procedure: Spinal Mobilization With Leg Movement — spinal mobilization with leg movement is the intervention given to experimental group. This technique involves applying pressure to the relevant spinous process while the patient moves their limb through the previously restricted range of motion. It is assumed that the restriction of movement is due to a spinal issue but it does not always indicate nerve damage as spinal movement is necessary for limb movement beyond a certain point. The goal is to address any spinal mechanical limitations and there may also be potential effects on the nerves.
  Arms: Group A
Procedure: Spinal Mobilization — The patients will be given Spinal mobilization transverse glide(kaltenborn glide) on the effected spinous process. The total time duration will be 25-30 minutes.
  Arms: Group B
Procedure: Conventional treatment — Participants will be given Hot pack for 15 minutes, TENS for 10 minutes

SUMMARY:
This study will be a Randomized Control Trial in which Both Genders with Age between 20 to 50 Years who had diagnosed with lumbar radiculopathy will be recriuted in to two groups.group A will be recieving spinal mobilzation with leg movement along with TENS & hot pack.whie group B will be given only spinal mobilization with TENS & hot pack.before and after the introduction of interventions pain,disabaility,speed of gait,cadence and SLR will be checked before and after the treatment

DETAILED DESCRIPTION:
Lumbar Radiculopathy is a medical condition that occurs when one or more nerve roots in the spinal cord are compressed or damaged, leading to pain, weakness, numbness or tingling sensations in the affected area of the body. This condition can be caused by herniated discs, spinal stenosis, Degenerative disc disease, tumors and infections.This study will be a Randomized Control Trial.The study will be conducted in district Swabi. We will recruit the data from NCS University Rehabilitation Centre Swabi.oswestry disbaility index will be given at the start of study and NPRS to check their pain and disbaility levels.SMWLM will be given to experimental group.Participants will be given Hot pack for 15 minutes, TENS for 10 minutes.The patient receives a set of three repetitions, then three sets of six repetitions, with a 30-second break in between each set of treatments. In this session, a progression was also provided as free SLR overpressure. A total of 6 sessions will be given thrice a week on alternate days for 2 consecutive weeks. The treatment will be given with 5 repetitions of SMWLM and 10 repetitions of spinal mobilization with three sets of transverse glide. Total time duration of the treatment will be around 25-35 minutes§ Pre assessment will be conducted at baseline followed by intervention for 3 days per week for 6 consecutive weeks.Final assessment will be conducted at the end of 6 weeks of intervention

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lumbar Radiculopathy with unilateral radiating leg pain.
* Both Genders with Age between 20 to 50 Years.
* Patient willing to participate and complete their follow-ups.
* Pain from (0-35 degrees) in Straight Leg Raise(Dural Pain).
* Positive neurodynamic test i.e. SLR test(35-70 degrees),which indicate sciatica)
* Pain more 3-5 or More on NPRS.

Exclusion Criteria:

* Spinal stenosis.
* Cauda equina syndrome.
* Patients having Somatic referred pain.
* Specific diseases of spine like ankylosing spondylitis, ,vertebral collapse, Rheumatoid arthritis, and Spondylolisthesis.
* Tb spine, intermittent claudication,diabetic neuropathy.
* Recent infection.
* Mental retardation.
* Previous spinal Surgery.
* Pelvis Fracture.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
pain severity | 2 weeks
  Pain will be measured using Numeric Pain Rating Scale which is an eleven point scale scored from 0 indicating no pain and 10 indicating worst pain

SECONDARY OUTCOMES:
Straight leg raise | 2 weeks
  Goniometer is a manual scale use for measuring the range of motion of a joint. In this scale degree varies from 0-360 angle
Lumbar Disability | 2 weeks
  Lumbar disability will be measured using Oswestry Disability Index which is a valid and reliable tool consisting of 10 items from which patient gets to choose according to their level of function
Cadence | 2 weeks
  10 METER WALK TEST: Initial 2 meters of the gait and final 2 meters of the gait will be for acceleration and deceleration. And the patient is then asking to walk and will assess the cadence and speed.

CONTACTS AND LOCATIONS:
Locations (1):
- NCS University Rehabilitaion Centre Swabi, Swabi, KPK, Pakistan